CLINICAL TRIAL: NCT02803463
Title: Peritoneal Closure Versus Non Closure During Open Appendectomy: a Randomized Trial
Brief Title: Peritoneal Closure Versus Non Closure During Open Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16_12_2015-23/14
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Acute Appendicitis
Keywords: peritoneal closure; appendectomy; postoperative pain; life quality
MeSH Terms: conditions — Appendicitis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peritoneal Closure (Active Comparator): open appendectomy with peritoneal closure
  Interventions: Procedure: open appendectomy with peritoneal closure
- Peritoneal Non Closure (Active Comparator): open appendectomy without peritoneal closure
  Interventions: Procedure: open appendectomy without peritoneal closure

INTERVENTIONS:
Procedure: open appendectomy with peritoneal closure — open appendectomy with peritoneal closure under general anesthesia for acute appendicitis
  Arms: Peritoneal Closure
Procedure: open appendectomy without peritoneal closure — open appendectomy without peritoneal closure under general anesthesia for acute appendicitis
  Arms: Peritoneal Non Closure

SUMMARY:
There has been no consensus over closure versus non closure of peritoneum during abdominal operations. The aim of this study is to compare the effect of peritoneal closure versus non closure over postoperative pain, early complications and life quality.

DETAILED DESCRIPTION:
There has been no consensus over closure versus non closure of peritoneum during abdominal operations. in literature, few reports suggested that peritoneal closure may prolong the operation time, may increase the costs and has a probable aggravating effect on postoperative pain. In addition, there have been some reports that suggest non closure of peritoneum may not increase the postoperative complications. The need of further studies to clarify the effect of peritoneal closure versus non closure on postoperative pain and life quality especially has been specified in some literature. The aim of this study is to compare the effect of peritoneal closure versus non closure over postoperative pain, early complications and life quality.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute appendicitis
* age between 18-65 years

Exclusion Criteria:

* preoperatively diagnosed intraabdominal abcess
* intraoperatively diagnosed free purulent fluid in abdominal cavity
* pregnancy
* malignancy history
* mental retardation
* chronical renal failure
* chronical liver disease
* diabetes mellitus
* patients' denial of participation to study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain score | postoperative day 1
  visual analogue score for pain at postoperative day 1 via using 10 cm vas scale.
Surgical Site Infection | postoperative 30 days
  Postoperative Surgical Site Infection in 30 days following surgery includes incisional infections and intrabdominal abcess
Life Quality Score | postoperative day 10
  Euro-Qol 5D-5L for assesment of life quality at postoperative day 10th

SECONDARY OUTCOMES:
operation time | intraoperatively
  time from beginning of incision to closure of incision
wound dehiscence | postoperative 30 days
  fascial dehiscence during postoperative 30 days diagnosed via physical examination of sonography.
postoperative mortality | postoperative 30 days
  mortality in postoperative 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin K Bektasoglu, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bektasoglu HK, Hasbahceci M, Yigman S, Yardimci E, Kunduz E, Malya FU. Nonclosure of the Peritoneum during Appendectomy May Cause Less Postoperative Pain: A Randomized, Double-Blind Study. Pain Res Manag. 2019 May 23;2019:9392780. doi: 10.1155/2019/9392780. eCollection 2019. PMID 31249637